CLINICAL TRIAL: NCT05785182
Title: Optical Coherence Tomography Imaging to Visualize Bacteria or Biofilm on Hardware, Bone and Soft Tissue in Open Fracture and Infected Fracture
Brief Title: OCT in Open Fracture and Infected Fracture
Status: Recruiting | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Dartmouth College (Other)
Responsible Party: Principal Investigator, Ida Leah Gitajn, Section Chief, Orthopaedics, Dartmouth-Hitchcock Medical Center
Other Study IDs: STUDY02001786
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Trauma Injury; Trauma; Open Fracture; Fracture Infection
MeSH Terms: conditions — Accidental Injuries; Wounds and Injuries; Fractures, Open | interventions — Open Fracture Reduction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Open Fracture: High energy open fracture.
  Interventions: Procedure: Open Fracture
- Infected Fracture: Infected open or closed fracture.
  Interventions: Procedure: Infected Fracture

INTERVENTIONS:
Procedure: Open Fracture — Patients 18 years of age or older with open fracture. Provision of informed consent.
  Groups: Open Fracture
Procedure: Infected Fracture — Patients 18 years of age or older with infected fracture. Provision of informed consent.
  Groups: Infected Fracture

SUMMARY:
This is a pilot prospective, observational study of patients with open or infected fracture evaluating the feasibility and acceptability of OCT, a light-based imaging modality that requires no drug or contrast agent.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Open fracture
* Fracture Related Infection

Exclusion Criteria:

* Metatarsal fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age or older who present to DHMC (Lebanon) with open and infected fracture
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility and acceptability of OCT imaging | 36 months
  The primary objective of this work is to demonstrate feasibility, acceptability, and preliminary effectiveness of Optical Coherence Tomography (OCT) to image bacteria and biofilm.
  Data will be analyzed accordingly: The association between optical imaging parameters (particularly around biofilm and bacterial contamination) and (1) surgical wound severity and (2) development of infection or treatment failure for infection.

CONTACTS AND LOCATIONS:
Overall Officials: Ida L Gitajn, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States